CLINICAL TRIAL: NCT02588716
Title: Effects of Terlipressin on Blood Loss and Transfusion Requirements During Major Liver Resection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, Lecturer, of Anesthesia & ICU, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Terlipressin
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2015-07

CONDITIONS: Hepatectomy, Surgical Blood Loss, Terlipressin
Keywords: Hepatectomy, Surgical Blood Loss, terlipressin
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Terlipressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terlipressin (Active Comparator): Terlipressin will be given at the beginning of surgery as an initial bolus dose of (1 mg over 30 mins) followed by a continuous infusion of 2μg/kg/h to be continued throughout the surgery then gradually withdrawn over 4 hours
  Interventions: Drug: Terlipressin
- Control (Placebo Comparator): same volumes of normal saline with the same rate of infusion, throughout the operation then gradually withdrawn over 4 hours.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Terlipressin — Terlipressin will be given as an intravenous injection of 2μg/kg/h to be continued throughout the surgery and weaned off over four hours postoperatively.
  Other Names: glipressin
  Arms: Terlipressin
Drug: normal saline — Same volumes of normal saline infusion, throughout the operation then gradually withdrawn over 4 hours.
  Arms: Control

SUMMARY:
To evaluate the effects of Terlipressin infusion on blood loss & transfusion requirements in cirrhotic patients undergoing major liver resections.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age, American Society of Anesthesiology (ASA) classification class I and II and assigned for elective resection of 2 or more liver segments portal hypertension

Exclusion Criteria:

* Patients with Child-Turcotte-Pugh grade B or C, clinically significant portal hypertension (splenomegaly, thrombocytopenia with platelets < 1011/L, esophageal varices grade 2 or more), Preoperative renal failure (GFR < 50ml/min), heart failure, Bradyarrhythmia (heart rate < 60/min), history of hemorrhagic stroke, Uncontrolled arterial hypertension (Blood pressure >160/100mmHg), and Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
blood loss | intraoperative period
  blood loss in ml

SECONDARY OUTCOMES:
blood units transfused | intraoperative period
  number of packed RBCs units transfused
lactate level | at start and end of resection
  lactate level in blood gas sample in mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Derived] Abbas MS, Mohamed KS, Ibraheim OA, Taha AM, Ibraheem TM, Fadel BA, Elawamy A, Abbas AM. Effects of terlipressin infusion on blood loss and transfusion needs during liver resection: A randomised trial. Acta Anaesthesiol Scand. 2019 Jan;63(1):34-39. doi: 10.1111/aas.13226. Epub 2018 Aug 5. PMID 30079635